CLINICAL TRIAL: NCT04455191
Title: Comparison of the Effects of Thawing Embryos in Advance and Thawing on the Day of Transfer on Pregnancy Outcomes in the Frozen Embryo Transfer Cycle
Brief Title: Comparison of Thawing Embryos in Advance and on the Day of Transfer on Pregnancy Outcomes in FET Cycle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jinan Central Hospital (Other)
Responsible Party: Principal Investigator, Bin Wu, Reproductive medicine department, Jinan Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: JianCH-RM2020-001
Record Dates: First submitted 2020-06-28; First posted 2020-07-02 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: In Vitro Fertilization; Frozen Embryo Transfer
Keywords: Frozen embryos; Thawing

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thawing Embryos in Advance (Experimental): Thawing embryos one day in advance (16:00), 18h before embryos transfer (10:00).
  Interventions: Procedure: Thawing Embryos in Advance
- Thawing Embryos on the Day of Transfer (Experimental): Thawing embryos on the day of transfer (8:00), 2h before embryos transfer (10:00).
  Interventions: Procedure: Thawing Embryos on the Day of Transfer

INTERVENTIONS:
Procedure: Thawing Embryos in Advance — Thaw Embryos one day in Advance
  Arms: Thawing Embryos in Advance
Procedure: Thawing Embryos on the Day of Transfer — Thaw Embryos on the morning of transfer day.
  Arms: Thawing Embryos on the Day of Transfer

SUMMARY:
Respectively for patients with repeated transplant failure and routine patients, Thawing frozen embryos in advance (18h) to extend the duration of embryonic development or thawing embryos on the day of transfer in the frozen embryo transfer cycle, to analyze which way can improve clinical pregnancy outcomes, is there a significant difference between the two ways or two types of patients?

DETAILED DESCRIPTION:
Although in clinical practice, thawed embryos with appropriate development time will be selected strictly according to the number of days after ovulation, there are still two problems in actual clinical treatment: one is the embryonic factor, although the rate of embryonic development is generally the same, However, the phenomenon of delayed embryo division and development often occurs. The second is the endometrial factor. There are reports that a small number of people will move the transplant window forward, or the transplant window is narrow. This potentially creates the risk of embryo-endometrial mismatch. Based on this, the research team focused on patients with frozen embryo transfer cycles and put forward the strategy of "thawing embryos in advance and prolonging the development period of embryos properly" in an effort to achieve better repair of damage caused by embryo freezing and fine-tuning of embryo-endometrial interaction time. Therefore, it is necessary to compare thawing embryos in advance and thawing on the day of transfer on pregnancy outcomes in patients with repeated transplant failure and routine patients respectively.

The purpose of this study is to analyze which way can improve clinical pregnancy and birth outcomes, is there a significant difference between the two ways or two types of patients?

ELIGIBILITY:
Inclusion Criteria:

* Aged <=35 years old;
* Regular menstrual cycle;
* Baseline follicle stimulating hormone (FSH) <12 IU/L;
* Infertility, pure fallopian tube or/and male factor;
* At least 2 high-quality day 3 embryos or 1 high-quality day 5 blastocyst are used for ET.

Exclusion Criteria:

* Patients with repeated transplant failure:
* Abnormal uterus, such as adenomyosis, endometriosis, endometrial polyps or Asherman syndrome;
* Abnormal ovaries, such as low ovarian response and polycystic ovary syndrome (PCOS);
* The endometrial thickness of FET day is <7 mm.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women in childbearing age intend to do IVF-FET
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate (Pregnancy or Not) | 6 weeks
  Observe the clinical pregnancy rate under different embryo thawing time
Live Birth Rate (Birth or Not) | 40 weeks
  Observe the live birth rate under different embryo thawing time

CONTACTS AND LOCATIONS:
Overall Officials: Yingchun Zhang, Dr, Study Director — Jinan Central Hospital
Locations (1):
- Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong, China